CLINICAL TRIAL: NCT03794895
Title: Assessment of Efficacy of Uterine Artery Doppler in Predicting the Response to Mefenamic Acid During Treatment of Women With IUCD Associated Menorrhagia
Brief Title: Prediction of Response to IUCD Associated Menorrhagia Using Doppler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasmine Essam Eldin Mohamed Mohamed Ismail, Principal investigator, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Yasmine's Protocol
Record Dates: First submitted 2018-12-27; First posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Women's Health: Amenorrhea/Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Echocardiography, Doppler

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm clinical trial (Experimental)
  Interventions: Device: Doppler

INTERVENTIONS:
Device: Doppler — Doing doppler for women having IUCD associated menorrhagia

SUMMARY:
Studying the efficacy of uterine artery doppler in predicting response to mefenamic acid in women having IUCD associated menorrhagia

ELIGIBILITY:
Inclusion Criteria:

* women in chile bearing period (age 20-35 yrs ) with history of regular menstrual cycle presenting with recent onset of more then three months menorrhagia after IUCD "copper T 380 A" insertion

Exclusion Criteria:

* history of bleeding tendency
* history of abnormal uterine bleeding due to other causes
* history of active liver disease
* history of antiplatelet or anticoagulant intake in the last month
* history of thyroid disease
* history of endometritis
* history of allergy to NSAIDs
* Adenomyosis
* women having contraindications to use NSAIDs e.g. peptic ulcer
* Insulin dependant diabetes mellitus

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female having menorrhagia due to IUCD
Enrollment: 156 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Resistance index and Pulsitality index (Predicting the response to IUCD associated menorrhagia) | 1 year
  Base line uterine artery doppler is done to the patient complaining of IUCD related menorrhagia prior to treatment , parameters of doppler are: resistance index and pulsitality index, then the patient takes mefenamic acid tablets 500 mg three times daily for five days, assessment of response whether the patient is responder or not is done using pictorial blood loss assessment chart then base line doppler parameters in responders and non responders are compared to correlate the response to base line doppler parameters

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine Es Ismail, Bachelor, Principal Investigator — Ain Shams University
Locations (1):
- AinshamsU, Cairo, Abbaseya, Egypt